CLINICAL TRIAL: NCT00407316
Title: Quality of Life and Visual Function in Uveitis Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The New York Eye & Ear Infirmary (Other)
Other Study IDs: 07-A-6803
Record Dates: First submitted 2006-12-02; First posted 2006-12-05 (Estimated); Last update posted 2006-12-05 (Estimated); Status verified 2006-12

CONDITIONS: Anterior Uveitis; Posterior Uveitis; Panuveitis; Uveitis
Keywords: Uveitis; Quality of life; Visual function
MeSH Terms: conditions — Uveitis, Anterior; Uveitis, Posterior; Panuveitis; Uveitis

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The purpose of this study was to measure the quality of visual function and quality of daily living in patients with anterior, posterior, and panuveitis.

DETAILED DESCRIPTION:
The National Eye Institute Visual Functioning Questionnaire, version August 2000 (NEI VFQ-25) and the Medical Outcomes Study (MOS) 36 Item Short Form Health Survey Instrument (SF-36) (RAND 36-Item Health Survey 1.0 Questionnaire) will be administered by a trained interviewer. Socio-demographic and clinical data will be collected for additional QOL parameter.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent
* Subjects of either gender
* Age greater than or equal to 18 years of age
* Diagnosed with Uveitis

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2006-06; Study Completion 2006-11

CONTACTS AND LOCATIONS:
Overall Officials: C. Michael Samson, MD, Principal Investigator — New York Eye and Ear Infirmary
Locations (1):
- New York Eye and Ear Infirmary, New York, New York, United States